CLINICAL TRIAL: NCT04519177
Title: Randomized Trial of a Sleep Disorders Program on Firefighter Safety and Disability
Brief Title: Randomized Trial of a Sleep Disorders Program on Firefighter Safety and Disability ...
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Laura K. Barger, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 2020P002448
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Early Education) (Experimental): Firefighters in station randomized to the experimental (early education) will receive the sleep health education program (SHEP) including screening for common sleep disorders. Those found at high risk will be given information about seeking further evaluation, diagnosis and treatment, if necessary.
  Interventions: Behavioral: Sleep Health Education Program (SHEP)
- Control (Later education) (No Intervention): Firefighters in station randomized to the control condition will not receive SHEP prior to the data collection.

INTERVENTIONS:
Behavioral: Sleep Health Education Program (SHEP) — Sleep Health Education Program (SHEP) including screening for common sleep disorders
  Arms: Experimental (Early Education)

SUMMARY:
The investigators have shown that sleep health education and sleep disorders screening improve health and safety of employees. There is potential to increase the benefits of the sleep health education and screening program if more firefighters are evaluated, diagnosed and referred for treatment. Investigators will evaluate whether firefighters in stations randomized to participate in the Sleep Health and Education Program (SHEP) intervention will have improved health and safety outcomes as compared to firefighters in stations randomized to the control condition.

ELIGIBILITY:
Inclusion Criteria:

* Firefighters working in one of the two fire departments selected for study

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of sleep disorder | 12 months (on end-of-year questionnaire)
  Evaluation of sleep disorder
Diagnosis of sleep disorder | 12 months (on end-of-year questionnaire)
  Diagnosis of sleep disorder
Treatment of sleep disorder | 12 months (on end-of-year questionnaire)
  Treatment of sleep disorder
Injuries | Over 12 months (The number of injuries as documented in the fire department database)
  Injuries
Disability days | Over 12 months (The number of injuries as documented in the fire department database)
  Disability days

SECONDARY OUTCOMES:
Motor vehicle crashes | Over 12 months, reported on monthly surveys
  Motor vehicle crashes (exploratory aim)
Near crashes | Over 12 months, reported on monthly surveys
  Near crashes (exploratory aim)

IPD SHARING:
Plan to Share IPD: Yes
Results derived from the proposed work will be shared through presentation at research conferences as well as publication in peer-reviewed journals. We or the journal will submit an electronic version of all final manuscripts upon acceptance for publication to PubMed Central database, in compliance with NIH Policy. If required, published data will also be deposited in publicly available databases.
  Per NIH Policy, we will make the database available to other investigators following publication of the final study results. The database will not contain identifying information per HIPAA regulations and permission will be obtained from participants to share their data with researchers outside the BWH.
  Per Partners policies, any investigator or entity requesting the data must request the data in writing in an agreement outlining how the data will be used, protected, and maintained.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of results.
Access Criteria: Per the NIH Policy on Data Sharing, we will make the database available to other investigators following publication of the final study results. The database will not contain identifying information per the regulations outlined in HIPPA, and permission will be obtained from study participants to share their data with researchers outside the Brigham and Women's Hospital. Per Partners HealthCare System policies, any investigator or entity requesting the data must request the data in writing in an agreement outlining how the data will be used, protected, and maintained, e.g., through a formal Data Use Agreement (DUA) negotiated by a Partners office or a template letter agreement signed by the sharing and receiving PIs.